CLINICAL TRIAL: NCT06260254
Title: Effects of Railway Vibration on Sleep and Disease
Acronym: BioVib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: University of Pennsylvania (Other); University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 244826201
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Noise Exposure; Sleep Disturbance; Sleep Hygiene; Metabolic Disturbance; Cognitive Change; Glucose Metabolism Disorders (Including Diabetes Mellitus); Vibration; Exposure
Keywords: neurobehavioral performance; Traffic noise; auditory fatigue; polysomnography; metabolomics; vibration
MeSH Terms: conditions — Parasomnias; Sleep Hygiene; Glucose Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: All participants will be exposed to each of the different vibration conditions. Each study night is treated as a separate arm of the crossover study. The order of the vibration exposure conditions will be be randomly assigned across participants using a Latin square design to avoid first-order carryover effects. Each subject will be exposed to one night of each of the following:
  Quiet night: No noise or vibration will be played, serving as a control night to assess individual baseline sleep, metabolic profile, and cognitive performance; Three railway vibration nights to determine consequences of noise-disrupted sleep. The vibration level in these three nights will be 0.5 mm/s, 0.7 mm/s and 0.9 mm/s respectively, so that exposure-response relationships can be derived.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be aware that in any given study night they can be exposed to railway vibration and noise. They will not be informed what exposure condition will occur in any given night, but they can become unblinded to the exposure if they are awake, as they will may hear the noise or feel the vibration.
  Study investigators responsible for analysing cognitive performance variables and physiological sleep data will be be blind to which vibration and noise interventions were introduced on which study nights.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Night (No Intervention): Single study night with no noise exposure, to determine normal baseline sleep.
- Low Vibration Night (Experimental): Single study night with railway vibration and noise events, to determine consequences of sleep disturbance by railway vibration at a lower level
  Interventions: Radiation: Railway noise; Radiation: Low level railway vibration
- Intermediate Vibration Night (Experimental): Single study night with railway vibration and noise events, to determine consequences of sleep disturbance by railway vibration at an intermediate level
  Interventions: Radiation: Railway noise; Radiation: Intermediate level railway vibration
- High Vibration Night (Experimental): Single study night with railway vibration and noise events, to determine consequences of sleep disturbance by railway vibration at a higher level
  Interventions: Radiation: Railway noise; Radiation: High level railway vibration

INTERVENTIONS:
Radiation: Railway noise — Low level railway noise, not exceeding 50 dB LAF,max. Thirty six single railway noise events.
  Arms: High Vibration Night; Intermediate Vibration Night; Low Vibration Night
Radiation: Low level railway vibration — 36 single railway noise events at 0.5 mm/s, varying from 11.5 s to 56.9 s in duration. Vibration always occurs concurrently with the noise exposure.
  Arms: Low Vibration Night
Radiation: Intermediate level railway vibration — 36 single railway noise events at 0.7 mm/s, varying from 11.5 s to 56.9 s in duration. Vibration always occurs concurrently with the noise exposure.
  Arms: Intermediate Vibration Night
Radiation: High level railway vibration — 36 single railway noise events at 0.9 mm/s, varying from 11.5 s to 56.9 s in duration. Vibration always occurs concurrently with the noise exposure.
  Arms: High Vibration Night

SUMMARY:
This study will investigate the biological mechanisms linking sleep disruption by vibration and noise, and the development of cardiometabolic disease. In a laboratory sleep study, the investigators will play railway vibration of different levels during the night. The investigators will also measure objective sleep quality and quantity, cognitive performance across multiple domains, self-reported sleep and wellbeing outcomes, and blood samples. Blood samples will be analyzed to identify metabolic changes and indicators of diabetes risk in different nights. Identifying biomarkers that are impacted by sleep fragmentation will establish the currently unclear pathways by which railway vibration exposure at night can lead to the development of diseases in the long term, especially metabolic disorders including diabetes.

DETAILED DESCRIPTION:
The experimental sleep study has the overarching goal of deepening understanding of sleep disruption by railway vibration and noise and changes in cardiometabolic and cognitive function. To this end, the study will address the following study aim:

Aim 1: Determine the biological and neurobehavioral consequences of sleep disruption by railway vibration. The investigators will measure the sleep of healthy volunteers, and each morning will obtain blood samples for metabolomics metabolic function analysis and administer a neurocognitive test battery. The investigators will compare effects on sleep, metabolomics, metabolic function and cognitive function between quiet nights and nights with railway traffic vibration and noise. Dose-response relationships will be determined by comparing nights with different levels of vibration.

This study will take place in the sound environment laboratory (SEL) at the University of Gothenburg Department of Occupational and Environmental Medicine. The SEL is a high fidelity research laboratory equipped to simulate a typical apartment, including three individually light-, sound- and vibration-isolated private bedrooms. Ceiling mounted speakers in each room and electrodynamic transducers mounted to the underside of each bed allow the investigators to create a realistic acoustic environment by transmitting sound and vibration exposures from the control room to each bedroom individually. The investigators have shown previously that results from this lab with high ecological validity are comparable with results from the field.

This study has a prospective within-subjects cross-over design. Participants (total N=24) will each spend five consecutive nights in the SEL, with a sleep opportunity between 23:00-07:00. Daytime sleep will be prohibited, confirmed with measures of daytime activity via wrist actigraphy monitors worn continuously throughout the study. Three subjects will take part concurrently, in separate bedrooms. The first night is a habituation period to the study protocol and for familiarization with the test procedures. The second night will be a quiet condition without noise or vibration, to determine normal baseline sleep, cardiometabolic profile, and cognitive performance. Study nights 3-5 are the vibration nights and will be randomly assigned across participants using a Latin square design to avoid first-order carryover effects. In these vibration nights, vibration and noise from railway freight will be played into the bedrooms to determine the effects of vibration and noise on sleep, cardiometabolic function and cognitive performance. Thirty six trains will occur each night, randomly distributed across the 8-hour sleep period.

For railway vibration the investigators will use synthesized signals based on measured data, used in previous laboratory studies. It is necessary to use synthesized vibration, rather than recorded signals, so that the investigators can accurately adjust the acoustical character of the exposure as needed. Railway vibration will be accompanied by high fidelity recordings of railway freight noise. This is to maximize ecological validity of the exposures since vibration rarely occurs without noise, and to mask any mechanical sounds from the vibration transducers.

Vibration and noise exposures will reflect realistic railway freight traffic noise levels that occur in dwellings alongside railway lines in Sweden. The maximum Wm-weighted vibration amplitudes in the three vibration nights will be 0.5 mm/s, 0.7 mm/s and 0.9 mm/s respectively. Maximum sound pressure levels of individual train passages will not exceed 49.8 dB LAF,max. Trains will vary from 11.5 s to 56.9 s in duration. All vibration amplitudes will be calibrated on the mattress of the bed, under a 75 kg reference weight to simulate the bed being occupied. All sound pressure levels will be calibrated to 10 cm above the pillow in each bedroom prior to the study, so that these levels accurately reflect the noise exposure of the subjects during sleep.

Each night the investigators will record physiologic sleep with polysomnography (PSG) and cardiac activity with electrocardiography (ECG). Each study morning, subjects will provide a 2ml blood sample and answer questionnaires and will depart the SEL to follow their normal daytime routine. They will return to the SEL at 20:00 each evening to prepare for sleep measurements. Caffeine will be prohibited after 15:00 and alcohol will be prohibited at all times. Because extreme and/or variable dietary behavior can affect the metabolome/lipoprotein profile, participants will be given guidance that they should eat a similar evening meal on each day of the laboratory study, confirmed with a food diary. The actual meal itself can be different for different study participants, because the study has a within-subjects design.

Sleep will be recorded with ambulatory polysomnography (PSG) and cardiac activity with electrocardiography (ECG) and finger pulse photoplethysmogram. Data are recorded offline onto the sleep recorder, and will be downloaded and checked every study morning to ensure data quality. In addition to traditional sleep analysis, raw PSG data will be used to calculate the Odds Ratio Project, a novel metric of sleep depth and stability.

Each study morning subjects will provide a 2 ml blood sample for plasma metabolomics analysis. To ensure reliable data, blood samples will be taken at the same time every day to mitigate circadian effects, before eating or drinking anything except water, and each sample will be handled in the same way i.e. centrifuged, aliquoted and stored in -80C freezers. Subjects will eat the same food each study evening to mitigate within-subject dietary effects on the blood metabolome. Furthermore, a 2-hour oral glucose tolerance test (OGTT) will be performed in the mornings after the quiet control night (i.e. after study night 2) and after the third vibration exposure night (i.e. after study night 5). The investigators will measure response to a 75g glucose bolus at timepoints 10, 20, 30, 60, 90 and 120 minutes after the glucose administration.

Each evening, subjects will complete a computerized cognitive test battery taking approximately 20 minutes, that includes 10 tests across a range of cognitive domains (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance). Cognition data will be analyzed to determine key measures of cognitive speed and accuracy, adjusting for practice effects and the difficulty of the stimulus set.

Subjects will complete a battery of one-time validated questionnaires to measure their general health (SF-36), chronotype, noise sensitivity, habitual sleep quality, environmental sensitivity, and annoyance and sleep disturbance by noise. Subjects will also answer a questionnaire each study evening and morning, involving questions on sleepiness (Karolinska Sleepiness Scale), auditory fatigue, sleep disturbance by noise, and validated sleep and disturbance questions.

ELIGIBILITY:
Inclusion Criteria:

1) live in or around the city of Gothenburg area (Sweden)

Exclusion Criteria:

1. aged <18 or >30 years;
2. habitual sleep and wake timings more than ±1 hour different from the study sleep times (i.e. habitual sleep time should be 22:00-00:00 and habitual wake time should be 06:00-08:00);
3. BMI>25 kg/m2;
4. regular sleep medication use (prescribed or "over-the-counter");
5. poor hearing acuity (measured during screening via pure tone audiometry);
6. diagnosed with sleep disorders;
7. diagnosed with diabetes
8. indications of sleep apnea on the STOP-BANG questionnaire;
9. shift work;
10. smoking, vaping, snus, or other nicotine use;
11. pregnant or breastfeeding

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Fasting insulin resistance in the morning immediately after the Control night | One night
  Calculated using the Homeostatic model of insulin resistance (HOMA-IR)
Fasting insulin resistance in the morning immediately after the low vibration night | One night
  Calculated using the Homeostatic model of insulin resistance (HOMA-IR)
Fasting insulin resistance in the morning immediately after the intermediate vibration night | One night
  Calculated using the Homeostatic model of insulin resistance (HOMA-IR)
Fasting insulin resistance in the morning immediately after the high vibration night | One night
  Calculated using the Homeostatic model of insulin resistance (HOMA-IR)
Total sleep time during the Control night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total sleep time during the low vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total sleep time during the intermediate vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total sleep time during the high vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N1 sleep during the Control night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N2 sleep during the Control night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N3 sleep during the Control night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of rapid eye movement (REM) sleep during the Control night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N1 sleep during the low vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N2 sleep during the low vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N3 sleep during the low vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of rapid eye movement (REM) sleep during the low vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N1 sleep during the intermediate vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N2 sleep during the intermediate vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N3 sleep during the intermediate vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of rapid eye movement (REM) sleep during the intermediate vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N1 sleep during the high vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N2 sleep during the high vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N3 sleep during the high vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of rapid eye movement (REM) sleep during the high vibration night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Wakefulness after sleep onset (WASO) during the Control night | One night
  Total number of minutes awake during the night after the first appearance of sleep of any stage. Measured via Polysomnography /EEG, scored according to American Academy of Sleep Medicine guidelines.
Wakefulness after sleep onset (WASO) during the low vibration night | One night
  Total number of minutes awake during the night after the first appearance of sleep of any stage. Measured via Polysomnography /EEG, scored according to American Academy of Sleep Medicine guidelines.
Wakefulness after sleep onset (WASO) during the intermediate night | One night
  Total number of minutes awake during the night after the first appearance of sleep of any stage. Measured via Polysomnography /EEG, scored according to American Academy of Sleep Medicine guidelines.
Wakefulness after sleep onset (WASO) during the high vibration night | One night
  Total number of minutes awake during the night after the first appearance of sleep of any stage. Measured via Polysomnography /EEG, scored according to American Academy of Sleep Medicine guidelines.
Number of awakenings during the Control night | One night
  Measured via Polysomnography /EEG, scored according to American Academy of Sleep Medicine guidelines.
Number of awakenings during exposure to low vibration | One night
  Measured via Polysomnography /EEG, scored according to American Academy of Sleep Medicine guidelines.
Number of awakenings during exposure to intermediate vibration | One night
  Measured via Polysomnography /EEG, scored according to American Academy of Sleep Medicine guidelines.
Number of awakenings during exposure to high vibration | One night
  Measured via Polysomnography /EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep onset latency (SOL) during the Control Night | One night
  Defined as the time from lights out to the first epoch of sleep. Measured via Polysomnography /EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep onset latency (SOL) during the low vibration night | One night
  Defined as the time from lights out to the first epoch of sleep. Measured via Polysomnography /EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep onset latency (SOL) during the intermediate vibration night | One night
  Defined as the time from lights out to the first epoch of sleep. Measured via Polysomnography /EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep onset latency (SOL) during the high vibration night | One night
  Defined as the time from lights out to the first epoch of sleep. Measured via Polysomnography /EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep efficiency during the Control night | One night
  Defined as the percentage of time in bed spent in a non-wake sleep stage, measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep efficiency during the low vibration night | One night
  Defined as the percentage of time in bed spent in a non-wake sleep stage, measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep efficiency during the intermediate vibration night | One night
  Defined as the percentage of time in bed spent in a non-wake sleep stage, measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
S Sleep efficiency during the high vibration night | One night
  Defined as the percentage of time in bed spent in a non-wake sleep stage, measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep depth assessed using the odds ratio product (ORP) during the Control night | One night
  Average ORP over the full night, from 0 (never occurs during wake) to 2.5 (only occurs during wake). Derived via polysomnography/EEG measurements.
Sleep depth assessed using the odds ratio product (ORP) during the low vibration night | One night
  Average ORP over the full night, from 0 (never occurs during wake) to 2.5 (only occurs during wake). Derived via polysomnography/EEG measurements.
Sleep depth assessed using the odds ratio product (ORP) during the intermediate vibration night | One night
  Average ORP over the full night, from 0 (never occurs during wake) to 2.5 (only occurs during wake). Derived via polysomnography/EEG measurements.
Sleep depth assessed using the odds ratio product (ORP) during the high vibration night | One night
  Average ORP over the full night, from 0 (never occurs during wake) to 2.5 (only occurs during wake). Derived via polysomnography/EEG measurements.
Maximal change of odds ratio product (ORP) during exposure to railway vibration events | One night
  Measure of acute sleep disruption by noise, calculated as the difference between the ORP in the 30s prior to noise onset and the maximum ORP during railway vibration. Averaged over 36 vibration events during the night.
Area under the curve of odds ratio product (ORP) during exposure to railway vibration events, calculated using the trapezoid rule | One night
  Measure of acute sleep disruption by noise, calculated as the difference between the ORP in the 30s prior to noise onset and the maximum ORP during railway vibration. Averaged over 36 vibration events during the night.
N-acetylglucosamine/galactosamine (GlycA) concentration after the Control night | One night
  Determined from NMR analysis of blood plasma
N-acetylglucosamine/galactosamine (GlycA) concentration after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
N-acetylglucosamine/galactosamine (GlycA) concentration after exposure to intermediate vibration | One night
  Determined from NMR analysis of blood plasma
N-acetylglucosamine/galactosamine (GlycA) concentration after exposure to high vibration | One night
  Determined from NMR analysis of blood plasma
Sialic acid (GlycB) concentration after the Control night | One night
  Determined from NMR analysis of blood plasma
Sialic acid (GlycB) concentration after exposure to low vibration | One night
  Determined from NMR analysis of blood plasma
Sialic acid (GlycB) concentration after exposure to intermediate vibration | One night
  Determined from NMR analysis of blood plasma
Sialic acid (GlycB) concentration after exposure to high vibration | One night
  Determined from NMR analysis of blood plasma
Supramolecular phospholipid composite (SPC) concentration after the Control night | One night
  Determined from NMR analysis of blood plasma
Supramolecular phospholipid composite (SPC) concentration after exposure to low vibration | One night
  Determined from NMR analysis of blood plasma
Supramolecular phospholipid composite (SPC) concentration after exposure to intermediate vibration | One night
  Determined from NMR analysis of blood plasma
Supramolecular phospholipid composite (SPC) concentration after exposure to high vibration | One night
  Determined from NMR analysis of blood plasma
Ethanol concentration (mmol/L) after the Control night | One night
  Determined from NMR analysis of blood plasma
Ethanol concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Ethanol concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Ethanol concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Trimethylamine-N-oxide concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Trimethylamine-N-oxide concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Trimethylamine-N-oxide concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Trimethylamine-N-oxide concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
2-Aminobutyric acid concentration (mmol/L) after exposure to Control night | One
  Determined from NMR analysis of blood plasma
2-Aminobutyric acid concentration (mmol/L) after exposure to low vibration night | One
  Determined from NMR analysis of blood plasma
2-Aminobutyric acid concentration (mmol/L) after exposure to intermediate vibration night | One
  Determined from NMR analysis of blood plasma
2-Aminobutyric acid concentration (mmol/L) after exposure to high vibration night | One
  Determined from NMR analysis of blood plasma
Alanine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Alanine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Alanine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Alanine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Asparagine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Asparagine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Asparagine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Asparagine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Creatine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Creatine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Creatine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Creatine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Creatinine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Creatinine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Creatinine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Creatinine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Glutamic acid concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Glutamic acid concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Glutamic acid concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Glutamic acid concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Glutamine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Glutamine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Glutamine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Glutamine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Glycine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Glycine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Glycine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Glycine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Histidine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Histidine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Histidine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Histidine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Isoleucine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Isoleucine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Isoleucine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Isoleucine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Leucine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Leucine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Leucine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Leucine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Lysine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Lysine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Lysine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Lysine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Methionine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Methionine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Methionine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Methionine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
N,N-Dimethylglycine concentration (mmol/L) after Control night | One night
  Determined from NMR analysis of blood plasma
N,N-Dimethylglycine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
N,N-Dimethylglycine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
N,N-Dimethylglycine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Ornithine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Ornithine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Ornithine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Ornithine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Phenylalanine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Phenylalanine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Phenylalanine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Phenylalanine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Proline concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Proline concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Proline concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Proline concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Sarcosine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Sarcosine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Sarcosine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Sarcosine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Threonine concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Threonine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Threonine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Threonine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Tyrosine concentration (mmol/L) after exposure toControl night | One night
  Determined from NMR analysis of blood plasma
Tyrosine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Tyrosine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Tyrosine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Valine concentration (mmol/L) after Control night | One night
  Determined from NMR analysis of blood plasma
Valine concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Valine concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Valine concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
2-Hydroxybutyric acid concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
2-Hydroxybutyric acid concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
2-Hydroxybutyric acid concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
2-Hydroxybutyric acid concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Acetic acid concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Acetic acid concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Acetic acid concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Acetic acid concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Citric acid concentration (mmol/L) after Control night | One night
  Determined from NMR analysis of blood plasma
Citric acid concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Citric acid concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Citric acid concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Formic acid concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Formic acid concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Formic acid concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Formic acid concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Lactic acid concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Lactic acid concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Lactic acid concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Lactic acid concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Succinic acid concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Succinic acid concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Succinic acid concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Succinic acid concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Choline concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Choline concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Choline concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Choline concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
2-Oxoglutaric acid concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
2-Oxoglutaric acid concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
2-Oxoglutaric acid concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
2-Oxoglutaric acid concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
3-Hydroxybutyric acid concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
3-Hydroxybutyric acid concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
3-Hydroxybutyric acid concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
3-Hydroxybutyric acid concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Acetoacetic acid concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Acetoacetic acid concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Acetoacetic acid concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Acetoacetic acid concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Acetone concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Acetone concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Acetone concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Acetone concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Pyruvic acid concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Pyruvic acid concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Pyruvic acid concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Pyruvic acid concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
D-Galactose concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
D-Galactose concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
D-Galactose concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
D-Galactose concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Glucose concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Glucose concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Glucose concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Glucose concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Glycerol concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Glycerol concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Glycerol concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Glycerol concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Dimethylsulfone concentration (mmol/L) after exposure to Control night | One night
  Determined from NMR analysis of blood plasma
Dimethylsulfone concentration (mmol/L) after exposure to low vibration night | One night
  Determined from NMR analysis of blood plasma
Dimethylsulfone concentration (mmol/L) after exposure to intermediate vibration night | One night
  Determined from NMR analysis of blood plasma
Dimethylsulfone concentration (mmol/L) after exposure to high vibration night | One night
  Determined from NMR analysis of blood plasma
Response to an oral glucose bolus, calculated as area under curve for glucose, in the morning after the control night | One night
  Area under the curve (AUC) calculated using the trapezoidal rule, from glucose samples collected 10, 20, 30, 60, 90 and 120 minutes after the glucose bolus.
Response to an oral glucose bolus, calculated as area under curve for glucose, in the morning after the low vibration night | One night
  Area under the curve (AUC) calculated using the trapezoidal rule, from glucose samples collected 10, 20, 30, 60, 90 and 120 minutes after the glucose bolus.
Response to an oral glucose bolus, calculated as area under curve for glucose, in the morning after the intermediate vibration night | One night
  Area under the curve (AUC) calculated using the trapezoidal rule, from glucose samples collected 10, 20, 30, 60, 90 and 120 minutes after the glucose bolus.
Response to an oral glucose bolus, calculated as area under curve for glucose, in the morning after the high vibration night | One night
  Area under the curve (AUC) calculated using the trapezoidal rule, from glucose samples collected 10, 20, 30, 60, 90 and 120 minutes after the glucose bolus.
Response to an oral glucose load calculated as area under curve for insulin, in the morning after the low vibration night | One night
  Area under the curve (AUC) calculated using the trapezoidal rule, from insulin samples collected 10, 20, 30, 60, 90 and 120 minutes after the glucose bolus
Response to an oral glucose load calculated as area under curve for insulin, in the morning after the intermediate vibration night | One night
  Area under the curve (AUC) calculated using the trapezoidal rule, from insulin samples collected 10, 20, 30, 60, 90 and 120 minutes after the glucose bolus
Response to an oral glucose load calculated as area under curve for insulin, in the morning after the high vibration night | One night
  Area under the curve (AUC) calculated using the trapezoidal rule, from insulin samples collected 10, 20, 30, 60, 90 and 120 minutes after the glucose bolus
Early response to an oral glucose load calculated as area under curve for insulin, in the morning after the control night | One night
  Area under the curve (AUC) calculated using the trapezoidal rule, from insulin samples collected 10, 20 and 30 minutes after the glucose bolus
Early response to an oral glucose load calculated as area under curve for insulin, in the morning after the low vibration night | One night
  Area under the curve (AUC) calculated using the trapezoidal rule, from insulin samples collected 10, 20 and 30 minutes after the glucose bolus
Early response to an oral glucose load calculated as area under curve for insulin, in the morning after the intermediate vibration night | One night
  Area under the curve (AUC) calculated using the trapezoidal rule, from insulin samples collected 10, 20 and 30 minutes after the glucose bolus
Early response to an oral glucose load calculated as area under curve for insulin, in the morning after the high vibration night | One night
  Area under the curve (AUC) calculated using the trapezoidal rule, from insulin samples collected 10, 20 and 30 minutes after the glucose bolus
Glucose tolerance in the morning after exposure to low vibration, assessed as glucose concentration 120 minutes after a glucose bolus | One night
  Glucose concentrations determined from plasma samples with the Hexokinase/G-6-PDH method
Glucose tolerance in the morning after exposure to intermediate vibration, assessed as glucose concentration 120 minutes after a glucose bolus | One night
  Glucose concentrations determined from plasma samples with the Hexokinase/G-6-PDH method
Glucose tolerance in the morning after exposure to high vibration, assessed as glucose concentration 120 minutes after a glucose bolus | One night
  Glucose concentrations determined from plasma samples with the Hexokinase/G-6-PDH method
Glucose tolerance in the morning after Control night, assessed as glucose concentration 120 minutes after a glucose bolus | One night
  Glucose concentrations determined from plasma samples with the Hexokinase/G-6-PDH method
Stumvoll Insulin sensitivity Index in the morning after control | One night
  .226 - 0.0032 × BMI - 0.0000645 × I120 - 0.00375 × G90, where I120 and G90 represent insulin concentration 120 minutes after the glucose bolus, and glucose concentration 90 minutes after the glucose bolus, respectively.
Stumvoll Insulin sensitivity Index in the morning after exposure to low vibration | One night
  .226 - 0.0032 × BMI - 0.0000645 × I120 - 0.00375 × G90, where I120 and G90 represent insulin concentration 120 minutes after the glucose bolus, and glucose concentration 90 minutes after the glucose bolus, respectively.
Stumvoll Insulin sensitivity Index in the morning after exposure to intermediate vibration | One night
  .226 - 0.0032 × BMI - 0.0000645 × I120 - 0.00375 × G90, where I120 and G90 represent insulin concentration 120 minutes after the glucose bolus, and glucose concentration 90 minutes after the glucose bolus, respectively.
Stumvoll Insulin sensitivity Index in the morning after exposure to high vibration | One night
  .226 - 0.0032 × BMI - 0.0000645 × I120 - 0.00375 × G90, where I120 and G90 represent insulin concentration 120 minutes after the glucose bolus, and glucose concentration 90 minutes after the glucose bolus, respectively.
Matsuda insulin sensitivity index in the morning after control exposure | One night
  Calculated as 10,000/square root of [fasting glucose × fasting insulin] × [mean glucose × mean insulin during oral glucose tolerance test])
Matsuda insulin sensitivity index in the morning after exposure to low vibration | One night
  Calculated as 10,000/square root of [fasting glucose × fasting insulin] × [mean glucose × mean insulin during oral glucose tolerance test])
Matsuda insulin sensitivity index in the morning after exposure to intermediate vibration | One night
  Calculated as 10,000/square root of [fasting glucose × fasting insulin] × [mean glucose × mean insulin during oral glucose tolerance test])
Matsuda insulin sensitivity index in the morning after exposure to high vibration | One night
  Calculated as 10,000/square root of [fasting glucose × fasting insulin] × [mean glucose × mean insulin during oral glucose tolerance test])

SECONDARY OUTCOMES:
Evening subjective sleepiness, assessed using the Karolinska Sleepiness Scale after exposure to control | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Evening subjective sleepiness, assessed using the Karolinska Sleepiness Scale after exposure to low vibration | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Evening subjective sleepiness, assessed using the Karolinska Sleepiness Scale after exposure to intermediate vibration | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Evening subjective sleepiness, assessed using the Karolinska Sleepiness Scale after exposure to high vibration | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Morning subjective sleepiness, assessed using the Karolinska Sleepiness Scale after exposure to control | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Morning subjective sleepiness, assessed using the Karolinska Sleepiness Scale after exposure to low vibration | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Morning subjective sleepiness, assessed using the Karolinska Sleepiness Scale after exposure to intermediate vibration | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Morning subjective sleepiness, assessed using the Karolinska Sleepiness Scale after exposure to high vibration | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Self-reported sleep disturbance by vibration after control exposure | One night
  Assessed on a 0-10 numerical scale, from "Not at all" to "Extremely"
Self-reported sleep disturbance by vibration after exposure to low vibration | One night
  Assessed on a 0-10 numerical scale, from "Not at all" to "Extremely"
Self-reported sleep disturbance by vibration after exposure to intermediate vibration | One night
  Assessed on a 0-10 numerical scale, from "Not at all" to "Extremely"
Self-reported sleep disturbance by vibration after exposure to high vibration | One night
  Assessed on a 0-10 numerical scale, from "Not at all" to "Extremely"
Morning positive affect, assessed using the Positive and Negative Affect Schedule (PANAS) after control exposure | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Morning positive affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to low vibration | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Morning positive affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to intermediate vibration | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Morning positive affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to high vibration | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Morning negative affect, assessed using the Positive and Negative Affect Schedule (PANAS) after control exposure | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Morning negative affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to low vibration | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Morning negative affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to intermediate vibration | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Morning negative affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to high vibration | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Evening negative affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to control | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Evening negative affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to low vibration | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Evening negative affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to intermediate vibration | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Evening negative affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to high vibration | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Evening positive affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to control | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Evening positive affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to low vibration | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Evening positive affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to intermediate vibration | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Evening positive affect, assessed using the Positive and Negative Affect Schedule (PANAS) after exposure to high vibration | One night.
  PANAS is a 20-item instrument in which 20 words describing current mood and emotional state are rated on a 5-point Likert scale from "Not at all" to "Extremely". A composite positive affect score is calculated from 10 of these.
Event-related cardiovascular activation in response to control | One night
  Change in heart rate (ECG)
Event-related cardiovascular activation in response to low vibration | One night
  Change in heart rate (ECG)
Event-related cardiovascular activation in response to intermediate vibration | One night
  Change in heart rate (ECG)
Event-related cardiovascular activation in response to high vibration | One night
  Change in heart rate (ECG)
Evening neurobehavioural speed | One night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Evening neurobehavioural accuracy | One night
  Average of one key accuracy indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Smith, PhD, Principal Investigator — Göteborg University
Locations (1):
- University of Gothenburg, Gothenburg, Västra Götaland County, Sweden